CLINICAL TRIAL: NCT03155932
Title: An Open-label, Pilot, Proof of Concept Study to Evaluate the Safety, Tolerability, and Efficacy of Oral Etrasimod (APD334) in Patients With Primary Biliary Cholangitis
Brief Title: Safety, Tolerability, and Efficacy of Etrasimod (APD334) in Participants With Primary Biliary Cholangitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Arena Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APD334-010
Record Dates: First submitted 2017-05-11; First posted 2017-05-16 (Actual); Results first posted 2022-03-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-02

CONDITIONS: Primary Biliary Cholangitis
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — etrasimod

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- APD334 (Experimental): APD334 active treatment for 24 weeks.
  Interventions: Drug: APD334

INTERVENTIONS:
Drug: APD334 — APD334 active treatment for 24 weeks.
  Other Names: etrasimod

SUMMARY:
The purpose of this open-label, pilot, proof of concept study is to evaluate the safety, tolerability, and efficacy of oral etrasimod (APD334) in participants with primary biliary cholangitis (PBC).

ELIGIBILITY:
Key Inclusion Criteria:

* Males or females aged 18 to 80 years (inclusive) at the time of screening, with confirmed Primary Biliary Cholangitis (PBC) diagnosis based upon at least 2 of 3 criteria:

  * Anti-mitochondrial antibodies (AMA) titer >1:40 on immunofluorescence or M2 positive by enzyme-linked immunosorbent assay (ELISA) or positive PBC-specific antinuclear antibodies (anti-GP210 and/or anti-SP100)
  * Alkaline phosphatase (ALP) >1.5 x upper limit of normal (ULN) for at least 6 months
  * Liver biopsy findings consistent with PBC
* Use of ursodeoxycholic acid (UDCA) for at least 6 months prior to screening (stable dose for at least 3 months immediately prior to screening)
* Participants must have ALP >1.5 x ULN but <10 x ULN, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <5 x ULN, and total bilirubin <ULN, at all screening visits
* AST, ALT, ALP, and total bilirubin must have 2 values at least 4 weeks apart that are within 20% of each other

Key Exclusion Criteria:

* Chronic liver disease of a non-PBC etiology. However, PBC participants accompanied with primary Sjögren's syndrome (pSS) are eligible to be enrolled.
* History or evidence of clinically significant hepatic decompensation
* Medical conditions that may cause non-hepatic increases in ALP (e.g., Paget's disease)
* Clinically significant infections within 6 weeks prior to treatment start, or infection with hepatitis C virus anytime in the past
* Immunosuppressive, immunomodulating, or investigational agents within 30 days prior to treatment start
* Treatment with obeticholic acid (OCA) within 30 days prior to Day 1

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-12-29 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arena CT.gov Administrator, Study Director — Arena Pharmaceuticals
Locations (9):
- United States (4):
  - Gastroenterology and Hepatology, UC Davis Medical Center, Sacramento, California
  - Baylor College of Medicine, Houston, Texas
  - Texas Liver Institute, San Antonio, Texas
  - Swedish Medical Center, Seattle, Washington
- Australia (3):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Alfred Health, Melbourne, Victoria
- New Zealand (2):
  - Auckland City Hospital, Grafton, Auckland
  - Christchurch Clinical Studies Trust, Christchurch

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrollment was planned for up to 20 participants. Two participants were enrolled into the study and completed 24 weeks of treatment.
Groups:
- APD334: Participants received APD334 1 mg tablet once daily (qd) by mouth for 12 weeks. The dose for APD334 was escalated to 2 mg at Week 12 to Week 24, based on the participant's safety and pharmacokinetic (PK) data.
Period: Overall Study
Arm/Group | APD334
Started | 2
Participants Escalated to 2 mg Dose of APD334 at Week 12 to Week 24 | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | APD334
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — Reporting demographic results for this study in which only two participants were enrolled introduces the risk of participant identification. In order to protect the participant's privacy, results for the study cannot be reported.
  Male | NA — Reporting demographic results for this study in which only two participants were enrolled introduces the risk of participant identification. In order to protect the participant's privacy, results for the study cannot be reported.
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | NA — Reporting demographic results for this study in which only two participants were enrolled introduces the risk of participant identification. In order to protect the participant's privacy, results for the study cannot be reported.
  Asian | NA — Reporting demographic results for this study in which only two participants were enrolled introduces the risk of participant identification. In order to protect the participant's privacy, results for the study cannot be reported.
  Native Hawaiian or Other Pacific Islander | NA — Reporting demographic results for this study in which only two participants were enrolled introduces the risk of participant identification. In order to protect the participant's privacy, results for the study cannot be reported.
  Black or African American | NA — Reporting demographic results for this study in which only two participants were enrolled introduces the risk of participant identification. In order to protect the participant's privacy, results for the study cannot be reported.
  White | NA — Reporting demographic results for this study in which only two participants were enrolled introduces the risk of participant identification. In order to protect the participant's privacy, results for the study cannot be reported.
  More than one race | NA — Reporting demographic results for this study in which only two participants were enrolled introduces the risk of participant identification. In order to protect the participant's privacy, results for the study cannot be reported.
  Unknown or Not Reported | NA — Reporting demographic results for this study in which only two participants were enrolled introduces the risk of participant identification. In order to protect the participant's privacy, results for the study cannot be reported.

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum Alkaline Phosphatase (ALP) Concentration
Description: Reduction in ALP concentration is a surrogate marker of slower disease progression.
Time Frame: Baseline, Week 24
Population: Analyses were not conducted due to low enrollment (N=2). In order to protect participant's privacy, the results from the enrolled participants cannot be reported.
Arm/Group | APD334
Number analyzed (Participants) | 0

2. Primary Outcome: Number of Participants With Adverse Events
Description: Safety was assessed by monitoring adverse events and clinically relevant changes in vital signs and clinical laboratory results.
Time Frame: Up to Week 26
Population: Two participants who were enrolled and received treatment in this study.
Measure: Count of Participants; unit: Participants
Groups:
- APD334: Participants received APD334 1 mg tablet qd by mouth for 12 weeks. The dose for APD334 was escalated to 2 mg at Week 12 to Week 24, based on the participant's safety and PK data.
Arm/Group | APD334
Number analyzed (Participants) | 2
Participants | 2

3. Secondary Outcome: Change in Serum ALP Concentration
Description: Reduction in ALP concentration is a surrogate marker of slower disease progression.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Arm/Group | APD334
Number analyzed (Participants) | 0

4. Secondary Outcome: Pharmacokinetic Parameters of Etrasimod, and Its Metabolites
Time Frame: Up to Week 24
Population: as for outcome 1
Arm/Group | APD334
Number analyzed (Participants) | 0

5. Other Pre Specified Outcome: Exploratory - Change in Complete Blood Count
Time Frame: Baseline, Week 12, Week 24
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Exploratory - Change in Incidence of Fatigue as Assessed by Peripheral Biliary Cholangitis (PBC-40) Scale
Time Frame: Baseline, Week 12, Week 24
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Exploratory - Change in Incidence of Pruritus as Assessed by 5-Dimensions (5-D) Itch Scale
Time Frame: Baseline, Week 12, Week 24
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Exploratory - Change in Schirmer Test Outcome
Time Frame: Baseline, Week 12, Week 24
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Exploratory - Change in Tear Film Break-Up Time
Time Frame: Baseline, Week 12, Week 24
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Exploratory - Change in Concentration of Serum High Sensitivity C-Reactive Protein (hsCRP)
Time Frame: Baseline, Week 12, Week 24
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Exploratory - Change in Concentration of Serum Alanine Transaminase (ALT)
Time Frame: Baseline, Week 12, Week 24
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Exploratory - Change in Concentration of Serum Aspartate Transaminase (AST)
Time Frame: Baseline, Week 12, Week 24
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Exploratory - Change in Concentration of Serum Gamma-Glutamyl Transferase (GGT)
Time Frame: Baseline, Week 12, Week 24
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Exploratory - Change in Concentration of Serum C4
Time Frame: Baseline, Week 12, Week 24
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Exploratory - Change in Concentration of Serum Immunoglobulin
Time Frame: Baseline, Week 12, Week 24
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Exploratory - Change in Concentration of Serum GP73
Time Frame: Baseline, Week 12, Week 24
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Exploratory - Change in Concentration of Serum Anti-Mitochondrial Antibodies (AMA)
Time Frame: Baseline, Week 12, Week 24
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Exploratory - Change in Quality of Life
Time Frame: Baseline, Week 12, Week 24
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to Week 26
Description: A TEAE was defined as any adverse events (AE) that were reported following study treatment administration and up to 2 weeks after the last treatment intake. An SAE was any untoward medical occurrence that at any dose resulted in the following outcomes: death, was life-threatening, required/prolonged hospitalization, disability/incapacity, congenital anomaly/birth defect, and important medical events.
Arm/Group | APD334
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | APD334 (N=2)
Skin rash (Skin and subcutaneous tissue disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Worsening right hip pain (Musculoskeletal and connective tissue disorders) | 1
Elevated gamma-glutamyl transferase-worsening (Investigations) | 1
Loose stools (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Common cold - Upper respiratory tract infection (Infections and infestations) | 1
Elevated alkaline phosphatase-worsening (Investigations) | 1
Lower abdominal cramps (Gastrointestinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Cognitive defects (Nervous system disorders) | 1
Olecranon bursitis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-27): https://cdn.clinicaltrials.gov/large-docs/32/NCT03155932/Prot_SAP_001.pdf